CLINICAL TRIAL: NCT04878718
Title: Vancomycin and Fecal Microbiota Transplant in a Single Patient for the Treatment of Autism Spectrum Disorder
Brief Title: Vancomycin and Fecal Microbiota Transplant in a Single Patient With Autism Spectrum Disorder
Status: No longer available | Type: Expanded Access
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: 19343
Record Dates: First submitted 2021-04-28; First posted 2021-05-07 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Fecal Transplant
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Fecal Microbiota Transplantation; Vancomycin

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Fecal Microbiota Transplant; Vancomycin — Subject will be treated with vancomycin followed by fecal microbiota transplant
  Other Names: FMT; vancomycin

SUMMARY:
Single patient with ASD will be treated with Vancomycin followed by FMT.

DETAILED DESCRIPTION:
A single patient with profound ASD will be treated with Vancomycin. This will be followed by fecal microbiota transplant. The patient will be followed for one year.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Autism Spectrum Disorder
2. Parent or Legally Authorized Representative willing and able to provide informed consent
3. A reliable caregiver who can report side effects and communicate effectively with the research team
4. Stable medications in the two months prior to enrollment
5. Currently receiving interventions in the community/school for ASD
6. If female and of childbearing potential, must be willing to utilize at least one highly effective method of birth control for the duration of the study. This includes condoms with spermicide, oral birth control pills, contraceptive implants, intra-uterine devices, or diaphragms. Subjects not of reproductive potential will be exempt (e.g. post-menopausal, surgically sterilized)
7. If male, and partner is of childbearing potential, must be willing to utilize at least one highly effective method of birth control for the duration of the study. This includes condoms with spermicide, oral birth control pills, contraceptive implants, intra-uterine devices, or diaphragms. Subjects not of reproductive potential will be exempt (surgically sterilized)

Exclusion Criteria:

1. Female subjects who are pregnant, nursing, or intend to become pregnant during the study period.
2. Subjects whose caregivers are unable/unwilling to cooperate with the protocol requirements.
3. Subject will be excluded who are suffering with Rett syndrome and Childhood Disintegrative Disorder.
4. Other serious co-morbid medical disorders affecting brain function and behaviour, including uncontrolled seizures.
5. Subjects unable to refrain from taking non-study antibiotics for the period of the study.
6. Subjects diagnosed with cancer, except small localized basal cell carcinoma.
7. Subjects known to abuse alcohol or drugs.
8. Subjects who have undergone gastric bypass or total colectomy, or who are scheduled for these procedures.
9. Infection with HIV.
10. Infection with Hepatitis B or C.
11. Allergy to benzodiazepine.
12. Inability to stop loperamide, diphenoxylate/atropine, or cholestyramine before the study
13. Unable to stop opiate treatment unless on a stable dose including PRN dosing, and no dose increase planned for the duration of the study
14. Known positive stool cultures for enteropathogens including, but not limited to Shigella, Salmonella, and Campylobacter within 30 days before enrollment.
15. Known stool studies positive for ova and/or parasites in 30 days prior to enrollment.
16. Planned travel outside United States during study period.
17. Hypersensitivity to vancomycin
18. Renal insufficiency
19. Colitis

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Study Director — ProgenaBiome
Locations (1):
- Ventura Clinical Trials, Ventura, California, United States